CLINICAL TRIAL: NCT03919409
Title: A Randomized, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of TS-161 Administered Orally to Healthy Male and Female Participants
Brief Title: First-in-Human Study With Single and Multiple Doses of TS-161 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taisho Pharmaceutical R&D Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TS161-US101
Record Dates: First submitted 2019-04-15; First posted 2019-04-18 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Healthy Volunteers
Keywords: TS-161; CSF; first-in-human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Part A: Cohort 1: TS-161 15 mg (Experimental): Single dose of TS-161 15 mg or placebo in a fasted condition.
  Interventions: Drug: TS-161; Drug: TS-161 Placebo
- Part A: Cohort 2: TS-161 50 mg (Experimental): Single dose of TS-161 50 mg or placebo which will be dosed first in a fasted condition, and then in a fed condition, with a washout period in between 2 dosing. Although planned, all subsequent dose levels after Cohort 1 will be determined based on the results from the preceding cohorts.
  Interventions: Drug: TS-161; Drug: TS-161 Placebo
- Part A: Cohort 3: TS-161 100 mg (Experimental): Single dose of TS-161 100 mg or placebo in a fasted condition. Although planned, all subsequent dose levels after Cohort 1 will be determined based on the results from the preceding cohorts.
  Interventions: Drug: TS-161; Drug: TS-161 Placebo
- Part A: Cohort 4: TS-161 200 mg (Experimental): Single dose of TS-161 200 mg or placebo in a fasted condition. Although planned, all subsequent dose levels after Cohort 1 will be determined based on the results from the preceding cohorts.
  Interventions: Drug: TS-161; Drug: TS-161 Placebo
- Part A: Cohort 5: TS-161 400 mg (Experimental): Single dose of TS-161 400 mg or placebo in a fasted condition. Although planned, all subsequent dose levels after Cohort 1 will be determined based on the results from the preceding cohorts.
  Interventions: Drug: TS-161; Drug: TS-161 Placebo
- Part B: Cohort 6: TS-161 TBD (Experimental): Single dose of TS-161 in a fasted condition. The dose level will be determined based on the results from the preceding cohorts.
  Interventions: Drug: TS-161
- Part C: Cohort 7: TS-161 TBD (Experimental): Daily doses of TS-161 or placebo for 10 days in a fed condition. The dose level will be determined based on the results from the preceding cohorts.
  Interventions: Drug: TS-161; Drug: TS-161 Placebo
- Part C: Cohort 8: TS-161 TBD (Experimental): Daily doses of TS-161 or placebo for 10 days in a fed condition. The dose level will be determined based on the results from the preceding cohorts.
  Interventions: Drug: TS-161; Drug: TS-161 Placebo
- Part C: Cohort 9: TS-161 TBD (Experimental): Daily doses of TS-161 or placebo for 10 days in a fed condition. The dose level will be determined based on the results from the preceding cohorts.
  Interventions: Drug: TS-161; Drug: TS-161 Placebo

INTERVENTIONS:
Drug: TS-161 — TS-161 capsules
Drug: TS-161 Placebo — TS-161 matching placebo capsules
  Arms: Part A: Cohort 1: TS-161 15 mg; Part A: Cohort 2: TS-161 50 mg; Part A: Cohort 3: TS-161 100 mg; Part A: Cohort 4: TS-161 200 mg; Part A: Cohort 5: TS-161 400 mg; Part C: Cohort 7: TS-161 TBD; Part C: Cohort 8: TS-161 TBD; Part C: Cohort 9: TS-161 TBD

SUMMARY:
This is a Phase 1, first-in-human study involving single and multiple oral doses of TS-161 in healthy male and female participants. The safety, tolerability, pharmacokinetics and pharmacodynamics of TS-161 will be evaluated.

The study includes 3 parts; Part A (single ascending dose: Cohorts 1 to 5) , Part B (single dose, cerebrospinal fluid [CSF] collection: Cohort 6), and Part C (multiple ascending dose: Cohorts 7 to 9). Participants will be assigned to one of the 9 Cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult male and female participants between 18 and 55 years of age, inclusive
* Body weight ≥ 45 kg
* Body Mass Index (BMI) 18 - 30 kg/m^2, inclusive

Exclusion Criteria:

* Significant history or presence of medical disorders or condition capable of significantly affecting the absorption, metabolism, or elimination of drugs
* History or presence of psychiatric or neurologic disease or condition
* History of seizures
* Abnormal EEG observed at screening
* Abnormal blood pressure
* Breast cancer within the past 10 years, or any other malignancies within the past 5 years
* Clinically significant abnormal results in electrocardiogram, blood and urine test
* History or presence of liver disease
* Participants using medication or supplements within 14 days prior to dosing
* Use of N-methyl-D-aspartate (NMDA) receptor modulators (example: dextromethorphan, ketamine, amantadine, memantine) within 90 days of screening
* Loss of blood or blood products in excess of 450 mL within 60 days prior to screening
* Used any investigational drug within 60 days prior to screening
* Recent history of alcohol or drug abuse
* Any participant who currently uses or has used tobacco products or nicotine-containing products (cigarettes, pipes, e-cigarettes, nicotine patches, etc.) for one month or more prior to screening

Exclusion Criteria for Part B only:

* Significant abnormalities in lumbar spine
* History of clinically significant back pain, back pathology, and/or back injury
* History of migraines, and/or frequent, severe headaches
* History or presence of significant active bleeding or coagulation disorder or use of non-steroidal anti-inflammatory drugs or other drugs that affect coagulation or platelet function within 14 days prior to lumbar catheter insertion
* Allergy to lidocaine (Xylocaine®) or related drugs
* History of adverse reaction to lumbar puncture or epidural procedure

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2020-02-11 (Actual); Study Completion 2020-02-11 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of Adverse Events | Parts A and B: Day 1 to Day 8; Part C: Day 1 to Day 17
TS-161 Plasma Pharmacokinetic Profile - Cmax | Parts A and B: Day 1 predose and at multiple time points (up to 48 hours) postdose; Part C: Day 1 predose and at multiple time points (up to 12 hours) postdose, Day 2 to Day 9 predose, Day 10 predose and at multiple time points (up to 48 hours) postdose
  Maximum plasma concentration
TS-161 Plasma Pharmacokinetic Profile - Tmax | Parts A and B: Day 1 predose and at multiple time points (up to 48 hours) postdose; Part C: Day 1 predose and at multiple time points (up to 12 hours) postdose, Day 2 to Day 9 predose, Day 10 predose and at multiple time points (up to 48 hours) postdose
  Time to maximum plasma concentration
TS-161 Plasma Pharmacokinetic Profile - AUC(0-last) | Parts A and B: Day 1 predose and at multiple time points (up to 48 hours) postdose
  Area under the plasma concentration versus time curve from time zero to last measurable concentration
TS-161 Plasma Pharmacokinetic Profile - AUC(0-tau) | Part C: Day 1 predose and at multiple time points (up to 12 hours) postdose, Day 2 to Day 9 predose, Day 10 predose and at multiple time points (up to 48 hours) postdose
  Area under the plasma concentration versus time curve over a dosing interval
TS-161 Plasma Pharmacokinetic Profile - T1/2 | Parts A and B: Day 1 predose and at multiple time points (up to 48 hours) postdose; Part C: Day 1 predose and at multiple time points (up to 12 hours) postdose, Day 2 to Day 9 predose, Day 10 predose and at multiple time points (up to 48 hours) postdose
  Apparent terminal elimination half-life
TS-161 Plasma Pharmacokinetic Profile - CL/F | Parts A and B: Day 1 predose and at multiple time points (up to 48 hours) postdose; Part C: Day 1 predose and at multiple time points (up to 12 hours) postdose, Day 2 to Day 9 predose, Day 10 predose and at multiple time points (up to 48 hours) postdose
  Apparent clearance following oral administration
TS-161 Plasma Pharmacokinetic Profile - Vd,z/F | Parts A and B: Day 1 predose and at multiple time points (up to 48 hours) postdose; Part C: Day 1 predose and at multiple time points (up to 12 hours) postdose, Day 2 to Day 9 predose, Day 10 predose and at multiple time points (up to 48 hours) postdose
  Apparent volume of distribution following oral administration
TS-161 Urine Pharmacokinetic Profile - Ae | Part A: Day 1 predose and pooled for multiple intervals (up to 48 hours) postdose; Part C: Day 1 predose and pooled for multiple intervals (up to 48 hours after last dose) postdose
  Amount excreted in urine
TS-161 Urine Pharmacokinetic Profile - Fe% | Part A: Day 1 predose and pooled for multiple intervals (up to 48 hours) postdose; Part C: Day 1 predose and pooled for multiple intervals (up to 48 hours after last dose) postdose
  Percent of dose excreted in urine
TS-161 Urine Pharmacokinetic Profile - CLr | Part A: Day 1 predose and pooled for multiple intervals (up to 48 hours) postdose; Part C: Day 1 predose and pooled for multiple intervals (up to 48 hours after last dose) postdose
  Renal Clearance

SECONDARY OUTCOMES:
TS-161 CSF Pharmacokinetic Profile - Cmax | Part B: Day 1 predose and at multiple time points (up to 24 hours) postdose
  Maximum CSF concentration
TS-161 CSF Pharmacokinetic Profile - Tmax | Part B: Day 1 predose and at multiple time points (up to 24 hours) postdose
  Time to maximum CSF concentration
TS-161 CSF Pharmacokinetic Profile - AUC(0-last) | Part B: Day 1 predose and at multiple time points (up to 24 hours) postdose
  Area under the CSF concentration versus time curve from time zero to last
TS-161 CSF Pharmacokinetic Profile - T1/2 | Part B: Day 1 predose and at multiple time points (up to 24 hours) postdose
  Apparent terminal elimination half-life
Changes from baseline in relative and absolute powers of the delta, theta, alpha, beta and gamma bands using quantitative electroencephalogram (qEEG) compared to placebo | Part A: predose and at multiple time points (up to 8 hours) postdose

CONTACTS AND LOCATIONS:
Overall Officials: Taisho Director, Study Director — Taisho Pharmaceutical R&D Inc.
Locations (1):
- PAREXEL - Early Phase Clinical Unit-Los Angeles, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: No